CLINICAL TRIAL: NCT03858738
Title: A Prospective Pilot Study on Use of Liquid Crystal Contact Thermography to Detect Early Breast Cancer
Brief Title: A Pilot Study on Use of Liquid Crystal Contact Thermography to Detect Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: Braster S.A. (Industry)
Collaborators: Clinmark Clinical Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: ThermaAlg
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast pathology; malignancy; artificial intelligence; liquid crystal contact thermography; automatic algorithms; efficacy; sensitivity; specificity
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group A: women aged 25-49 years: Patient who had breast ultrasound done and classified according to the BI-RADS US classification, and the result was in category 4 or 5.
  Patient with indications for biopsy unless breast biopsy was performed in the last 3 months (except for FNA). Thermography examination was performed with the use of Braster device.
  Interventions: Device: Thermographic breast examination performed by Braster device
- Group B: Women aged 25-49 years or 50 ≥: Patient who had breast ultrasound done and classified according to the BI-RADS US classification, and the result was in category 1 or 2.Thermography examination was performed with the use of Braster device.
  Interventions: Device: Thermographic breast examination performed by Braster device
- Group C: Woman aged 50 years or over: Patient who had breast ultrasound done and classified according to the BI-RADS US classification, and the result was in category 4 or 5. Patient with indications for biopsy unless breast biopsy was performed in the last 3 months (except for FNA). Thermography examination was performed with the use of Braster device.
  Interventions: Device: Thermographic breast examination performed by Braster device

INTERVENTIONS:
Device: Thermographic breast examination performed by Braster device — Patient undergo contact thermography examination with the use of liquid crystal contact thermography device- Braster.
  Other Names: BRASTER™- IIa medical device, thermographic contact tester

SUMMARY:
The study was a multicentre, observational, cross-sectional, open and monitored trial involving 274 females who were subject to an examination using liquid crystal contact thermography device as a complementary tool to standard diagnostic imaging procedures of the breast glands. The study was conducted in specialist outpatient clinics. Patients were eligible to participate in the study upon signing the informed consent form. There was no follow up after the thermographic examination.

The study will comprise of a single registration of thermographic images of the breasts which will be subjected to automatic and expert analysis by radiologists.

ELIGIBILITY:
Inclusion Criteria:

Arm A:

1. Woman aged 25-49 years
2. Patient who had breast ultrasound done and classified according to the BI-RADS US classification, and the result was in category 4 or 5.
3. Patient with indications for biopsy unless breast biopsy was performed in the last 3 months (except for FNA).
4. Patient is able to read and understand the Patient Information Sheet and provided informed consent for participation in the study and disclosing medical data from the diagnostic process of the breast.

Arm B:

1. Woman aged 25-49 years or 50 years and above.
2. Patient who had breast ultrasound done and classified according to the BI-RADS US classification, and the result was in category 1 or 2.
3. Patient is able to read and understand the Patient Information Sheet and provided informed consent for participation in the study and disclosing medical data from the diagnostic process of the breast.

Arm C:

1. Woman aged 50 years or over.
2. Patient who had breast ultrasound done and classified according to the BI-RADS US classification, and the result was in category 4 or 5.
3. Patient with indications for biopsy unless breast biopsy was performed in the last 3 months (except for FNA).
4. Patient is able to read and understand the Patient Information Sheet and provided informed consent for participation in the study and disclosing medical data from the diagnostic process of the breast.

Exclusion Criteria:

For arms A and C

1. Patient after invasive diagnostic procedures of a breast lesion (a procedure performed less than 3 months prior to enrollment) - applies to CNB and MMT, does not apply to FNA.
2. Patient in the course of active infection with body temperature higher than 37.5°C.
3. Patient with symptomatic acute or chronic inflammation within the breast, visible signs of inflammation: pain, increased warmth, skin redness, oedema, breast abscesses, thrombosis.
4. Patient after trauma in the breast area with visible clinical signs of extravasation.
5. Patient in the course of oncological treatment for breast cancer.
6. Patient after breast surgery within 12 months prior to inclusion.
7. Patient with a history of conserving surgery for breast cancer (within 12 months after treatment).
8. Pregnant or breast-feeding patient.
9. Patient who consumed alcohol up to 2 hours before thermographic examination.
10. Patient after intense physical activity up to 30 minutes before thermographic examination.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women were eligible if they underwent a breast ultrasound (with outcome BIRADS 1-5), had no breast surgery over the previous year, no core biopsy over the previous 3 months, no previously-diagnosed breast cancer, were not pregnant or lactating, and had no symptoms/signs of local or generalized infection. Those recruited signed an informed consent form that also gave permission to use medical information (clinical characteristics, ultrasound, mammography and pathology findings) for study purposes. A total of 274 women, 25 years of age and older, were recruited consecutively between June 2015 and April 2016. Mammography was performed in some patients below 50 years and in all women of 50 years or over. The thermographic examination was performed after breast ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2016-06-08 (Actual); Study Completion 2016-08-19 (Actual)

PRIMARY OUTCOMES:
Diagnostic efficacy of liquid crystal contact thermography using a manual assessment algorithm as compared with ultrasound and/or mammography and breast biopsy. | 2 years
  C-statistic (area under receiver operator characteristic -ROC - curve) as measure of the ability of the thermographic findings to distinguish histologically-confirmed breast cancer from non-cancer, in women with abnormal breast ultrasound (BIRADS >3), stratified by age (<50 years; ≥50 years)